CLINICAL TRIAL: NCT07248943
Title: Contralateral Neural Tissue Mobilization for Cervical Radiculopathy: An Exploratory Study
Brief Title: Contralateral Neural Tissue Mobilization for Cervical Radiculopathy
Acronym: NTM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence In Motion (Other)
Collaborators: Rockhurst University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ContralateralNTM2025
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cervical Radiculopathy; Pain; Neuropathic Pain; Radicular Pain
Keywords: Cervical Radiculopathy; Neuropathic Pain; Peripheral Neuropathic Pain; Upper Extremity Pain; Radicular Pain; Cervical Spine Disorders; Nerve Root Compression; Neural Tissue Mobilization; Neurodynamic Mobilization; Neurodynamics; Contralateral Treatment; Median Nerve Mobilization; Upper Limb Neurodynamic Test (ULNT1a); Physical Therapy; Musculoskeletal Pain; Pain Phenotyping; Manual Therapy; Rehabilitation; Mechanosensitivity
MeSH Terms: conditions — Radiculopathy; Pain; Neuralgia; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Participants with unilateral cervical radiculopathy will receive a single treatment session of neural tissue mobilization applied to the contralateral (uninvolved) upper extremity. The intervention is delivered by licensed physical therapists with post-professional training in pain science and neurodynamic techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contralateral Neural Tissue Mobilization (Experimental): Participants with unilateral cervical radiculopathy will receive a single treatment session of neural tissue mobilization applied to the contralateral (uninvolved) upper extremity. The intervention is delivered by licensed physical therapists with post-professional training in pain science and neurodynamic techniques.
  Interventions: Behavioral: Contralateral Neural Tissue Mobilization (NTM)

INTERVENTIONS:
Behavioral: Contralateral Neural Tissue Mobilization (NTM) — A standardized 8-10 minute contralateral NTM protocol will be performed and includes:
  1. Supine passive neurodynamic mobilization (ULNT1a pattern) with:
     * Cervical side flexion toward the non-symptomatic side
     * Movement to the point of resistance
     * 1-2 seconds of gentle engagement followed by release
     * Repeated 15 times
  2. Supine passive neurodynamic mobilization with:
     * Neutral cervical position
     * Repeated 15 times
  3. Supine passive neurodynamic mobilization with:
     * Cervical side flexion away from the non-symptomatic side
     * Repeated 15 times
  4. Sitting active neurodynamic exercises (contralateral UE)
     * 10 active "sliders"
     * 10 active "tensioners"
     * 10 additional active "sliders" The neurodynamic pattern follows the ULNT1a sequence: shoulder abduction to 90°, external rotation, forearm supination, wrist/finger extension with ulnar deviation, and progressive elbow extension.
  Single treatment session delivered in-person by a trained physical therapist.

SUMMARY:
Cervical radiculopathy (CR) is a common form of peripheral neuropathic pain characterized by neck and upper extremity symptoms in a dermatomal distribution. Neural tissue mobilization (NTM) is an intervention shown to provide benefit for neuropathic pain presentations; however, some patients are unable to tolerate direct treatment of the symptomatic limb due to allodynia, hyperalgesia, or fear of movement. Early evidence from lower-extremity research suggests that contralateral NTM may produce therapeutic effects similar to ipsilateral treatment, but this approach has not been investigated in individuals with upper-extremity symptoms.

This exploratory case series aims to examine the immediate effects of contralateral NTM in adults presenting to outpatient physical therapy with CR. Participants will undergo pre- and post-treatment assessments of pain intensity, disability, fear-avoidance beliefs, pain distribution, and neurodynamic mechanosensitivity. Findings will provide preliminary evidence regarding whether contralateral NTM may serve as a viable treatment option when direct symptomatic limb treatment is not tolerated.

DETAILED DESCRIPTION:
Background and Rationale:

Pain phenotyping has emerged as an important clinical framework within physical therapy, enabling classification of pain presentations on the basis of pain mechanisms, clinical features, and patient-reported symptoms. Current pain phenotyping models identify three primary mechanisms: nociceptive, peripheral neuropathic, and nociplastic pain. Peripheral neuropathic pain is estimated to account for approximately one-quarter of patients presenting to outpatient physical therapy. It is characterized by pain arising from a lesion or disease of the somatosensory nervous system, with complex underlying biological mechanisms including neurogenic inflammation, immune dysregulation, demyelination, axonal loss, ion channel changes, and vascular alterations. Clinically, peripheral neuropathic pain commonly presents with pain in dermatomal or cutaneous nerve distributions, a history of nerve injury or mechanical compromise, and symptom provocation during neurodynamic or palpatory testing.

Cervical radiculopathy (CR) is a frequent and well-recognized form of peripheral neuropathic pain. CR most often results from intervertebral disc herniation or spondylosis, typically affecting the C7, C6, and C8 nerve roots. Patients commonly present with neck pain, upper extremity pain, and/or sensory, motor, or reflex deficits. Current evidence suggests that when patient presentation aligns with a peripheral neuropathic phenotype, interventions should be matched accordingly. Neural tissue mobilization (NTM) has demonstrated effectiveness in individuals with chronic neck and arm pain and is believed to exert beneficial effects through improvements in neuromeningeal mobility, blood flow, intraneural and extraneural fluid dynamics, inflammatory modulation, and graded exposure to movement.

However, some patients with CR present with significant allodynia, hyperalgesia, or fear of movement, making direct treatment of the symptomatic extremity challenging. Basic neuroanatomy and preliminary research suggest that contralateral NTM may produce therapeutic effects similar to ipsilateral NTM. Although early work in the lower extremity-including one clinical trial and one case study-has shown that contralateral NTM can reduce pain related to lumbar radiculopathy, this concept has not yet been explored in the upper extremity. Therefore, this exploratory study seeks to examine whether contralateral NTM produces immediate positive effects in patients presenting to physical therapy with CR.

Study Design:

This investigation uses a case-series design with pre- and post-intervention measures. A convenience sample will be recruited from four outpatient physical therapy clinics specializing in musculoskeletal pain. Clinicians participating in the study must have completed at least a 2-day (15-hour) post-professional training course in pain science and assessment of peripheral neuropathic pain, including instruction in NTM.

A total of approximately 40 patients aged 18 years or older will be recruited over a 3-month period. Eligible individuals must demonstrate unilateral arm pain in a dermatomal distribution consistent with CR, with or without neck pain. Exclusion criteria include bilateral upper-extremity pain, non-dermatomal pain, contraindications to NTM on the contralateral limb (e.g., recent surgery, significant tissue injury, allodynia), inability to read English, or unwillingness to consent.

Procedures and Outcome Measures:

After obtaining written informed consent, participants will complete baseline (pre-intervention) measures including:

Demographic questionnaire (non-identifiable data only)

Numeric Pain Rating Scale (NPRS) for upper-extremity pain

Neck Disability Index (NDI)

Fear-Avoidance Beliefs Questionnaire - Physical Activity subscale (FABQ-PA)

Pain drawing, quantified using a standardized grid overlay

Upper Limb Neurodynamic Test 1a (ULNT1a) of the affected limb, including goniometric measurement of elbow extension at symptom onset

Following baseline measures, each participant will receive a single treatment session of contralateral NTM, performed on the limb opposite the symptomatic side. The intervention consists of 8-10 minutes of standardized passive neurodynamic mobilizations in supine with specific variations in cervical positioning, followed by active "slider" and "tensioner" exercises in sitting.

Immediately after the intervention, participants will repeat all outcome measures (NPRS, FABQ-PA, pain drawing, and ULNT1a). After data collection is complete, clinical care will proceed according to the treating clinician's usual practice and will not be influenced by study procedures.

Data Handling and Analysis:

All data packets will be de-identified and coded by clinic and clinician. Data will be transferred to a secure electronic spreadsheet for analysis. Descriptive statistics (means, standard deviations, frequencies, and percentages) will summarize demographic variables and baseline characteristics. Pre- to post-intervention changes will be evaluated using paired t-tests with statistical significance set at p < 0.05.

Purpose of the Study:

The purpose of this exploratory case series is to determine whether contralateral neural tissue mobilization produces immediate changes in pain intensity, disability, fear-avoidance beliefs, pain distribution, and neurodynamic mechanosensitivity among individuals presenting with clinical features of cervical radiculopathy. Findings may inform future research and contribute to clinical understanding of whether contralateral NTM is a viable treatment option in patients unable to tolerate direct treatment of the symptomatic extremity

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older Presence of unilateral upper-extremity pain in a dermatomal distribution consistent with cervical radiculopathy (with or without neck pain)
* Able to read and understand English
* Willing and able to provide written informed consent
* New patient to the clinic or established patient who meets inclusion criteria and has not previously received neural tissue mobilization as part of treatment

Exclusion Criteria:

* Bilateral upper-extremity pain
* Upper-extremity pain that is non-dermatomal in distribution
* Presence of contraindications or precautions preventing use of the contralateral limb for neural tissue mobilization (e.g., injury, allodynia, recent surgery, postsurgical complications)
* Not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Pre-intervention to immediately post-intervention (same session).
  Change in patient-reported upper-extremity pain intensity measured using the 0-10 Numeric Pain Rating Scale, where 0 = no pain and 10 = worst imaginable pain. The NPRS is commonly used in musculoskeletal research to quantify pain severity.
Upper Limb Neurodynamic Test 1a (ULNT1a) - Elbow Extension Range | Pre-intervention to immediately post-intervention (same session).
  Change in degrees of elbow extension measured with a goniometer at the onset of symptoms during ULNT1a testing of the affected limb. The test assesses neurodynamic mechanosensitivity related to the median nerve.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Pre-intervention to immediately post-intervention (same session).
  Change in self-reported neck-related disability using the 10-item Neck Disability Index, scored from 0 to 50 and converted to a percentage (0-100%), with higher scores indicating greater disability.
Fear-Avoidance Beliefs Questionnaire - Physical Activity Subscale (FABQ-PA) | Pre-intervention to immediately post-intervention (same session).
  Change in fear-avoidance beliefs related to physical activity, assessed using the 4-item FABQ-PA (scores range from 0 to 24; higher scores indicate greater fear of physical activity).
Pain Drawing Area (Body Chart Grid Count) | Pre-intervention to immediately post-intervention (same session).
  Change in pain distribution quantified using a standardized body chart with an overlay grid. The number of grid blocks marked by the participant represents pain extent.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latimer J, Maher C, Refshauge K. The attitudes and beliefs of physiotherapy students to chronic back pain. Clin J Pain. 2004 Jan-Feb;20(1):45-50. doi: 10.1097/00002508-200401000-00009. PMID 14668656
- [Background] Gurudut P, Sherpa LB. Comparison of Ipsilateral Versus Contralateral LOwer Limb Neural Mobilization in Unilateral Lumbar Radiculopathy - A Randomized Clinical Trial. Int J Physiother. 2021;8(1):26-30.
- [Background] Louw A, Schmidt SG, Louw C, Puentedura EJ. Moving without moving: immediate management following lumbar spine surgery using a graded motor imagery approach: a case report. Physiother Theory Pract. 2015;31(7):509-17. doi: 10.3109/09593985.2015.1060656. PMID 26395828
- [Background] Gilbert KK, Smith MP, Sobczak S, James CR, Sizer PS, Brismee JM. Effects of lower limb neurodynamic mobilization on intraneural fluid dispersion of the fourth lumbar nerve root: an unembalmed cadaveric investigation. J Man Manip Ther. 2015 Dec;23(5):239-45. doi: 10.1179/2042618615Y.0000000009. PMID 26955255
- [Background] Song XJ, Gan Q, Cao JL, Wang ZB, Rupert RL. Spinal manipulation reduces pain and hyperalgesia after lumbar intervertebral foramen inflammation in the rat. J Manipulative Physiol Ther. 2006 Jan;29(1):5-13. doi: 10.1016/j.jmpt.2005.10.001. PMID 16396724
- [Background] Varangot-Reille C, Cuenca-Martinez F, Arribas-Romano A, Bertoletti-Rodriguez R, Gutierrez-Martin A, Mateo-Perrino F, Suso-Marti L, Blanco-Diaz M, Calatayud J, Casana J. Effectiveness of Neural Mobilization Techniques in the Management of Musculoskeletal Neck Disorders with Nerve-Related Symptoms: A Systematic Review and Meta-Analysis with a Mapping Report. Pain Med. 2022 Apr 8;23(4):707-732. doi: 10.1093/pm/pnab300. PMID 34633462
- [Background] Basson A, Olivier B, Ellis R, Coppieters M, Stewart A, Mudzi W. The Effectiveness of Neural Mobilization for Neuromusculoskeletal Conditions: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2017 Sep;47(9):593-615. doi: 10.2519/jospt.2017.7117. Epub 2017 Jul 13. PMID 28704626
- [Background] Tanaka N, Fujimoto Y, An HS, Ikuta Y, Yasuda M. The anatomic relation among the nerve roots, intervertebral foramina, and intervertebral discs of the cervical spine. Spine (Phila Pa 1976). 2000 Feb 1;25(3):286-91. doi: 10.1097/00007632-200002010-00005. PMID 10703098
- [Background] Murphy DR, Hurwitz EL, Gerrard JK, Clary R. Pain patterns and descriptions in patients with radicular pain: does the pain necessarily follow a specific dermatome? Chiropr Osteopat. 2009 Sep 21;17:9. doi: 10.1186/1746-1340-17-9. PMID 19772560
- [Background] Iyer S, Kim HJ. Cervical radiculopathy. Curr Rev Musculoskelet Med. 2016 Sep;9(3):272-80. doi: 10.1007/s12178-016-9349-4. PMID 27250042
- [Background] Smart KM, Blake C, Staines A, Thacker M, Doody C. Mechanisms-based classifications of musculoskeletal pain: part 2 of 3: symptoms and signs of peripheral neuropathic pain in patients with low back (+/- leg) pain. Man Ther. 2012 Aug;17(4):345-51. doi: 10.1016/j.math.2012.03.003. Epub 2012 Mar 31. PMID 22465002
- [Background] Schmid AB, Nee RJ, Coppieters MW. Reappraising entrapment neuropathies--mechanisms, diagnosis and management. Man Ther. 2013 Dec;18(6):449-57. doi: 10.1016/j.math.2013.07.006. Epub 2013 Sep 2. PMID 24008054
- [Background] Schmid AB, Fundaun J, Tampin B. Entrapment neuropathies: a contemporary approach to pathophysiology, clinical assessment, and management. Pain Rep. 2020 Jul 22;5(4):e829. doi: 10.1097/PR9.0000000000000829. eCollection 2020 Jul-Aug. PMID 32766466
- [Background] Kim KH, Moon SH, Hwang CJ, Cho YE. Prevalence of Neuropathic Pain in Patients Scheduled for Lumbar Spine Surgery: Nationwide, Multicenter, Prospective Study. Pain Physician. 2015 Sep-Oct;18(5):E889-97. PMID 26431142
- [Background] Orita S, Yamashita T, Ohtori S, Yonenobu K, Kawakami M, Taguchi T, Kikuchi SI, Ushida T, Konno SI, Nakamura M, Fujino K, Matsuda S, Yone K, Takahashi K. Prevalence and Location of Neuropathic Pain in Lumbar Spinal Disorders: Analysis of 1804 Consecutive Patients With Primary Lower Back Pain. Spine (Phila Pa 1976). 2016 Aug 1;41(15):1224-1231. doi: 10.1097/BRS.0000000000001553. PMID 26967122
- [Background] Cook, CE, DI Rhon, J Bialosky, M Donaldson, SZ George, T Hall, G Kawchuk, et al. 2023. "Developing Manual Therapy Frameworks for Dedicated Pain Mechanisms." Journal of Orthopaedic & Sports Physical Therapy (JOSPT) 1 (1): 48-62.
- [Background] Nijs J, Kosek E, Chiarotto A, Cook C, Danneels LA, Fernandez-de-Las-Penas C, Hodges PW, Koes B, Louw A, Ostelo R, Scholten-Peeters GGM, Sterling M, Alkassabi O, Alsobayel H, Beales D, Bilika P, Clark JR, De Baets L, Demoulin C, de Zoete RMJ, Elma O, Gutke A, Hanafi R, Hotz Boendermaker S, Huysmans E, Kapreli E, Lundberg M, Malfliet A, Meziat Filho N, Reis FJJ, Voogt L, Zimney K, Smeets R, Morlion B, de Vlam K, George SZ. Nociceptive, neuropathic, or nociplastic low back pain? The low back pain phenotyping (BACPAP) consortium's international and multidisciplinary consensus recommendations. Lancet Rheumatol. 2024 Mar;6(3):e178-e188. doi: 10.1016/S2665-9913(23)00324-7. Epub 2024 Feb 1. PMID 38310923
- [Background] Hodges PW, Sowa G, O'Neill C, Vo N, Foster N, Samartzis D, Lotz J. Development and application of predictive clinical biomarkers for low back pain care: recommendations from the ISSLS phenotype/precision spine focus group. Eur Spine J. 2025 Apr;34(4):1309-1318. doi: 10.1007/s00586-025-08720-4. Epub 2025 Feb 18. PMID 39964488